CLINICAL TRIAL: NCT00005239
Title: Genetic Epidemiology of Coronary Heart Disease Risk in Women Twins
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1120; R01HL041830 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2004-06

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases

SUMMARY:
To examine genetic and environmental influences on several recently identified coronary heart disease risk factors in identical and fraternal adult women twins. The risk factors included low density lipoprotein (LDL) subclass patterns, plasma apolipoprotein levels, body fat distribution, and serum insulin levels.

DETAILED DESCRIPTION:
BACKGROUND:

In 1974, a twin registry was established from members of the Kaiser Permanente Medical Care Program's Northern California region. In all, 9,821 twin pairs were enrolled. In 1978-1979, 434 pairs of female twins were recruited from the registry for a clinical examination of coronary heart disease risk factors. The clinical examination included an extensive health questionnaire, measurements of plasma lipids and serum chemistries, analyses of genetic markers for determination of zygosity, measurement of expired air carbon monoxide and serum thiocyanate levels, and a complete physical examination. During the ten years since the first examination, several new or more specific coronary heart disease risk factors have been recognized, including low density lipoprotein and insulin levels, and the anatomic distribution of body fat.

DESIGN NARRATIVE:

All women who participated in the first examination were invited to participate in the second examination. Medical records and/or death certificates were obtained to document coronary heart disease events. Questionnaires were used to collect information on health history, nutrition, and physical activity. A clinical examination assessed blood pressure, a variety of anthropometric measures and cardiovascular fitness. Blood specimens were collected for clinical chemistry and lipid/lipoprotein profiles. To assess genetic influence, the heritability of each of the risk factors was estimated. Blood was frozen for future studies of polymorphic DNA markers. Using the monozygotic co-twin control method, the effects of environmental or behavioral factors on these risk factors were assessed after controlling for genetic factors that could explain their association. Two hypotheses were examined that could be uniquely addressed using twin data. First, the association of body fat distribution with other coronary heart disease risk factors was mediated by serum insulin levels. Secondly, cardiovascular fitness explained in part the association of physical activity with coronary heart disease risk factors such as HDL-cholesterol and insulin levels. Lipoprotein analyses were conducted at Donner Laboratory at Berkeley.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1989-01; Study Completion 1991-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Selby — Kaiser Foundation Research Institute

REFERENCES:
- [Background] Austin MA, Sandholzer C, Selby JV, Newman B, Krauss RM, Utermann G. Lipoprotein(a) in women twins: heritability and relationship to apolipoprotein(a) phenotypes. Am J Hum Genet. 1992 Oct;51(4):829-40. PMID 1415225
- [Background] Edwards KL, Austin MA, Jarvik GP. Evidence for genetic influences on smoking in adult women twins. Clin Genet. 1995 May;47(5):236-44. doi: 10.1111/j.1399-0004.1995.tb04303.x. PMID 7554348
- [Background] Mayer EJ, Newman B, Quesenberry CP Jr, Selby JV. Usual dietary fat intake and insulin concentrations in healthy women twins. Diabetes Care. 1993 Nov;16(11):1459-69. doi: 10.2337/diacare.16.11.1459. PMID 8299435
- [Background] Austin MA, Hokanson JE. Epidemiology of triglycerides, small dense low-density lipoprotein, and lipoprotein(a) as risk factors for coronary heart disease. Med Clin North Am. 1994 Jan;78(1):99-115. doi: 10.1016/s0025-7125(16)30178-x. PMID 8283937
- [Background] Mayer EJ, Newman B, Quesenberry CP Jr, Friedman GD, Selby JV. Alcohol consumption and insulin concentrations. Role of insulin in associations of alcohol intake with high-density lipoprotein cholesterol and triglycerides. Circulation. 1993 Nov;88(5 Pt 1):2190-7. doi: 10.1161/01.cir.88.5.2190. PMID 8222114
- [Background] Selby JV, Austin MA, Newman B, Zhang D, Quesenberry CP Jr, Mayer EJ, Krauss RM. LDL subclass phenotypes and the insulin resistance syndrome in women. Circulation. 1993 Aug;88(2):381-7. doi: 10.1161/01.cir.88.2.381. PMID 8339401
- [Background] Austin MA, Newman B, Selby JV, Edwards K, Mayer EJ, Krauss RM. Genetics of LDL subclass phenotypes in women twins. Concordance, heritability, and commingling analysis. Arterioscler Thromb. 1993 May;13(5):687-95. doi: 10.1161/01.atv.13.5.687. PMID 8485120
- [Background] Edwards KL, Austin MA, Newman B, Mayer E, Krauss RM, Selby JV. Multivariate analysis of the insulin resistance syndrome in women. Arterioscler Thromb. 1994 Dec;14(12):1940-5. doi: 10.1161/01.atv.14.12.1940. PMID 7981183
- [Background] Selby JV, Austin MA, Sandholzer C, Quesenberry CP Jr, Zhang D, Mayer E, Utermann G. Environmental and behavioral influences on plasma lipoprotein(a) concentration in women twins. Prev Med. 1994 May;23(3):345-53. doi: 10.1006/pmed.1994.1048. PMID 8078856